CLINICAL TRIAL: NCT02349750
Title: Endometrial Scratch Injury Induced Higher Pregnancy Rate for Women With Unexplained Infertility Undergoing IUI With Ovarian Stimulation
Brief Title: Endometrial Scratch Injury in Women With Unexplained Infertility Undergoing IUI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, Assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 123
Record Dates: First submitted 2015-01-24; First posted 2015-01-29 (Estimated); Last update posted 2015-01-29 (Estimated); Status verified 2015-01

CONDITIONS: Unexplained Infertility
Keywords: Endometrial Scratch Injury; Unexplained infertility; intrauterine insemenation; ovulation induction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- endometrial scratch injury (Active Comparator): Patients received 100 mg of oral clomiphene citrate for five days starting on day 3 of the menstrual cycle, followed by daily injection of 150 IU of hMG and when more than two dominant follicles reached a diameter of 17 mm 5,000 IU of hCG was injected intramuscularly. Group S had ESI using No.8 neonatal feeding tube and after 24 to 36 hours, IUI was performed.
  Interventions: Procedure: endometrial scratch injury
- Non endometrial scratch injury (No Intervention): Patients received 100 mg of oral clomiphene citrate for five days starting on day 3 of the menstrual cycle, followed by daily injection of 150 IU of hMG and when more than two dominant follicles reached a diameter of 17 mm 5,000 IU of hCG was injected intramuscularly. Group C received IUI without ESI and after 24 to 36 hours, IUI was performed.

INTERVENTIONS:
Procedure: endometrial scratch injury — ESI using No.8 neonatal feeding tube
  Arms: endometrial scratch injury

SUMMARY:
The study included 154 infertile women Patients received 100 mg of oral clomiphene citrate for five days starting on day 3 of the menstrual cycle, followed by daily injection of 150 IU of hMG and when more than two dominant follicles reached a diameter of 17 mm 5,000 IU of hCG was injected intramuscularly. Patients were randomly allocated into two equal groups: Group C received IUI without ESI and Group S had ESI using No.8 neonatal feeding tube and after 24 to 36 hours, IUI was performed. Successful pregnancy was con-firmed by ultrasound and patients had failed trial underwent another trial of IUI for a maximum of three trials.

DETAILED DESCRIPTION:
The study included 154 infertile women with mean duration of infertility of 3.9±0.4 years. Patients received 100 mg of oral clomiphene citrate for five days starting on day 3 of the menstrual cycle, followed by daily injection of 150 IU of hMG and when more than two dominant follicles reached a diameter of 17 mm 5,000 IU of hCG was injected intramuscularly. Patients were randomly allocated into two equal groups: Group C received IUI without ESI and Group S had ESI using No.8 neonatal feeding tube and after 24 to 36 hours, IUI was performed. Successful pregnancy was con-firmed by ultrasound and patients had failed trial underwent another trial of IUI for a maximum of three trials.

ELIGIBILITY:
Inclusion Criteria:

1. Couple with unexplained infertility and assigned for IUI

Exclusion Criteria:

1. Woman's age of more than 40 years
2. Ovarian cyst detected in the ultrasound examination
3. Uterine lesions such as submucosal leiomyoma
4. A previous diagnosis of moderate to severe pelvic endometriosis
5. Women with body mass index ≥35 kg/m2 o
6. Women with signs of hyperandrogenemia dy

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 154 (Actual)
Dates: Start 2010-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
clinical pregnancy | 14 days after IUI

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Maged, MD, Principal Investigator — Kasr Alainy medical school